CLINICAL TRIAL: NCT01720979
Title: Attention, Learning and Behaviour Following Traumatic Brain Injury in Children
Brief Title: TBI Project Amsterdam
Status: Completed | Type: Observational
Sponsor: Marsh Königs (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor-Investigator, Marsh Königs, MSc, VU University of Amsterdam
Organization: VU University of Amsterdam (Other)
Other Study IDs: NL37226.029.11
Record Dates: First submitted 2012-10-25; First posted 2012-11-02 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Traumatic Brain Injury; Children; Prognosis; Neurocognition
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with traumatic injuries: Children that were admitted to the hospital after traumatic injuries to body parts below the clavicles (traumatic control injury) and children that were admitted to the hospital after traumatic brain injury as diagnosed by a physician (TBI).

SUMMARY:
Traumatic Brain Injury (TBI) is the world leading cause of acquired brain injury. Literature suggests a pivotal role for attentional functioning in neurocognitive and behavioural consequences of paediatric TBI. Limitations of traditional neuropsychological measures of attentional functioning have interfered with identification of the effect of paediatric TBI on attentional networks so far. Moreover, the associations between attentional networks, learning abilities, academic performance and behavioural and emotional problems following paediatric TBI are yet to be explored.

DETAILED DESCRIPTION:
Background:

Traumatic brain injury (TBI) is the world leading cause of disability in children (Winslade, 1998), causing deficits in motor function, neurocognition and adaptive behaviour (Anderson, 2001). Literature shows that age at injury is inversely related to the magnitude of deficits following TBI, highlighting the vulnerability of children for the effects of TBI.

The neurocognitive consequences of paediatric TBI have primarily been characterized by impairments in speed of information processing, attentional functioning and learning (Babikian & Asarnow, 2009; Catroppa & Anderson, 2009), interfering with typical neurocognitive development. We aim at elucidating the effects of TBI on neurocognitive function and investigate the relations between neurocognitive deficits, academic achievement and emotional and behavioural function, in order to improve our understanding of the post-injury functioning of children that have suffered TBI.

Methods:

Patients with TBI will be compared to a control group consisting of orthopedically injured patients. Orthopaedic control (OC) groups offer a better comparison to TBI patients than typically developing children by controlling for TBI risk factors related to neurocognition (e.g. Attention Deficit Hyperactivity Disorder, socioeconomic status), hospitalisation and the type of injuries other than brain injuries.

Measures:

Child's Orientation and Amnesia Test, Attention Network Test, Probabilistic Learning Test, Child Behaviour Checklist, Strengths & Difficulties Questionnaire, Experimental Neurocognitive Test developed at the VU University and Pupil Monitoring System.

ELIGIBILITY:
Inclusion Criteria:

TBI patients will be included if they

* have parental written informed consent
* provide written informed consent if aged over 11 years
* are Dutch speaking
* have a clinical diagnosis of TBI (closed head injury)
* have a time post-injury that is longer than 1 month
* are aged between 6-12 years.

Trauma control patients will be included if they:

* have parental written informed consent
* provide written consent if aged over 11 years
* are Dutch speaking
* have suffered an orthopaedic injury
* have no history of TBI
* and are aged between 6-12 years.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children that have been admitted to the hospital after sustaining trauma.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The white-matter integrity of children with TBI will be compared to children with traumatic control injuries | on average 1-year post-TBI
  FA/ADC values will be reported for selected region's of interest in children with TBI and children with traumatic control injuries.
Performance on tests of attention will be compared between children with TBI and children with traumatic control injuries | on average 1-year post-TBI
  Mean reaction time and accuracy will be reported for children with TBI and children with traumatic control injuries

SECONDARY OUTCOMES:
Parental reports of behavioural regulation will be compared between children with TBI and children with traumatic control injuries | on average 1-year post-TBI
  Problem scores on several types of behavioural problems will be reported for children with TBI and children with traumatic control injuries
Academic achievement will be compared between children with TBI and children with traumatic control injuries | on average 1-year post-TBI
  Scores on standardised tests of academic achievement will be reported for children with TBI and children with traumatic control injuries
Performance on test of reinforced learning will be compared between children with TBI and children with traumatic control injuries | on average 1-year post-TBI
  Reaction time and accuracy on computerised tests of reinforced learning will be reported for children with TBI and children with traumatic control injuries

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Oosterlaan, PhD, Principal Investigator — VU University of Amsterdam
Locations (5):
- Netherlands (5):
  - Libra rehabilitation centers Blixembosch Leijpark, Eindhoven - Tilburg, North Brabant
  - Academic Medical Center, Amsterdam, North Holland
  - VU University of Amsterdam, Amsterdam, North Holland
  - Merem revalidatiecentra de Trappenberg, Huizen, North Holland
  - Erasmus MC, Rotterdam, South Holland